CLINICAL TRIAL: NCT07100691
Title: Preoperative Metoclopramide to Enhance Gastric Emptying in Patients on Glucagon-Like Peptide-1 Receptor Agonists for Weight Loss: A Randomised Controlled Trial With Ultrasound Assessment
Brief Title: Gastric Emptying With Metoclopramide in GLP-1 Agonist Patients Undergoing Elective Surgery
Acronym: GEM-GLP1RA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Aneurin Moorthy, Consultant Anaesthesiologist, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEM-GLP1RA
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Aspiration During Anaesthetic Induction; Gastric Emptying Time; Preoperative Risk Assessment; Obesity (Disorder)
Keywords: GLP-1 Receptor Agonist; Metoclopramide; Elective Surgery; Residual Gastric Content; Gastric Ultrasound; Aspiration Risk; Perioperative Management; Obesity Medications; Randomised Controlled Trial; Anaesthesia Safety
MeSH Terms: conditions — Obesity | interventions — Metoclopramide

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to either standard care or standard care plus oral metoclopramide administered over 24 hours prior to surgery.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators performing and interpreting the ultrasound and collecting outcome data are blinded to group allocation. Patients are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants in this arm will continue their usual glucagon-like peptide-1 receptor agonist (GLP-1 RA) medication before surgery, in line with current perioperative guidance. No additional medications will be administered. Gastric ultrasound will be performed on the morning of surgery to assess residual gastric content.
- Metoclopramide + Standard Care (Experimental): Participants in this arm will continue their usual GLP-1 RA medication and also receive four oral doses of metoclopramide 10 mg: three doses the day before surgery and one dose on the morning of surgery. This intervention is intended to enhance gastric emptying and reduce residual gastric content, which will be assessed via gastric ultrasound on the morning of surgery.
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Metoclopramide — Oral metoclopramide 10 mg, administered as three doses the day before surgery and one dose on the morning of surgery (total four doses over 24 hours). Used to enhance gastric emptying in patients taking GLP-1 receptor agonists.
  Other Names: Maxolon
  Arms: Metoclopramide + Standard Care

SUMMARY:
This is a multicentre, investigator-blinded, randomised controlled trial evaluating whether the use of oral metoclopramide before surgery can reduce the amount of residual gastric content in patients who are taking glucagon-like peptide-1 receptor agonists (GLP-1 RAs) for weight loss. These medications are known to slow down gastric emptying, which may increase the risk of pulmonary aspiration during anaesthesia. Patients will be randomly assigned to either receive metoclopramide 24 hours before surgery or continue with standard care. The primary outcome will be the presence or absence of residual gastric content on ultrasound before surgery. Secondary outcomes include nausea, vomiting, constipation, and any adverse effects of the medication.

DETAILED DESCRIPTION:
The increasing use of glucagon-like peptide-1 receptor agonists (GLP-1 RAs) for weight loss has created a new challenge for anaesthesiologists: delayed gastric emptying in patients who appear to be fasted, which may increase their risk of pulmonary aspiration under anaesthesia. While consensus statements recommend assessing aspiration risk and implementing mitigation strategies, there is limited clinical trial evidence to support these practices.

This is a multicentre, prospective, single-blinded, randomised controlled trial designed to assess whether preoperative oral metoclopramide can reduce residual gastric content (RGC) in patients taking GLP-1 RAs prior to elective surgery. Eighty adult patients who are taking GLP-1 RAs for weight loss will be enrolled and randomly assigned in a 1:1 ratio to either standard care or standard care plus metoclopramide. Standard care is defined as continuation of GLP-1 RA medications as per current perioperative guidance. The intervention group will receive four doses of oral metoclopramide 10 mg: three doses the day before surgery and one dose on the morning of surgery.

The primary outcome for this randomised controlled trial will be the presence of residual gastric content (RGC) [yes/no] on gastric ultrasound examination in fasting patients taking GLP-1 agonists, scheduled for elective surgery. Our primary outcome will be a binary outcome, and we will define the presence of RGC as one or more of the following present on gastric ultrasound examination: 1. Presence of solid; 2. Presence thick fluid; and 3. > 1.5ml/kg of clear fluid.

Based on a recent published prospective cross-sectional study, the prevalence of increased RGC in patients taking GLP-1 agonist was 56% and the authors found that the absolute effect on RGC in patients taking GLP-1 agonists was 30% (i.e., increasing the chance of gastric contents by 30%) (11). Therefore, we propose that in the intervention group to reduce the prevalence of RGC to 25% to be clinically meaningful. Assuming Type 1 error = 0.05 and Type 2 error = 0.1 (80% power to detect this difference), then n= 36 patients will be required in each group. To accommodate for 10% participants who may withdraw from the study, we will aim to recruit n= 40 participants to each study arm, i.e. n=80 in total. Sample size calculation was verified using an online calculator (https://www.sealedenvelope.com/power/binary-superiority/)

Statistical analysis will be conducted on an intention-to-treat basis using appropriate tests for binary and continuous variables.

This trial aims to address the evidence gap in perioperative management of patients taking GLP-1 RAs and to evaluate whether a simple pharmacologic intervention with metoclopramide can safely reduce aspiration risk in this growing patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking GLP-1 receptor agonists (for weight loss only)
* Male and female patients aged 18 years or older
* Able to provide written informed consent
* ASA grade I-V
* Scheduled for elective surgery with an expected overnight hospital stay

Exclusion Criteria:

* Inability to provide informed consent
* Presence of hiatus hernia
* History of any gastric surgery
* Pregnancy
* Inability to lie in the right lateral decubitus position
* Patients taking chronic opioids
* Poorly controlled diabetes (HbA1c >69 mmol/mol)
* Urgent or emergency surgery, including trauma
* Diagnosis of Parkinson's disease
* Allergy or intolerance to metoclopramide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence of residual gastric content on preoperative gastric ultrasound | On the day of surgery prior to anaesthesia induction
  Residual gastric content (RGC) will be defined as the presence of any of the following on ultrasound prior to induction of anaesthesia: (1) solid content, (2) thick fluid, or (3) clear fluid >1.5 mL/kg in the gastric antrum. Ultrasound will be performed in the supine and right lateral decubitus positions by a blinded anaesthesiologist and reviewed by a second blinded assessor.

SECONDARY OUTCOMES:
Nausea/vomiting in PACU | 2 hours
  Nausea/Vomiting
Nausea/vomiting | 24 hours
  Nausea/vomiting
Constipation | 24 hours
  Constipation
Adverse Reactions to Metoclopramide | From enrollment to postoperative day 1.
  Adverse Reactions to Metoclopramide
Aspiration event | From the induction of anaesthesia to post-operative 6 hours
  Aspiration of gastric contents

CONTACTS AND LOCATIONS:
Overall Officials: Aneurin Moorthy, Principal Investigator — NOHC
Locations (2):
- Ireland (2):
  - National Orthopaedic Hospital Cappagh, Dublin, Dublin 5
  - Rotunda Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the limited scale of the study, the absence of an established data-sharing infrastructure, and institutional constraints regarding the release of health-related data beyond the study team. Any future sharing of anonymized data will require separate ethical approval and data access agreements.

REFERENCES:
- [Background] Perlas AK, R. POCUS Spotlight: Gastric Ultrasound. ASRA News. 2021;46.
- [Background] Sen S, Potnuru PP, Hernandez N, Goehl C, Praestholm C, Sridhar S, Nwokolo OO. Glucagon-Like Peptide-1 Receptor Agonist Use and Residual Gastric Content Before Anesthesia. JAMA Surg. 2024 Jun 1;159(6):660-667. doi: 10.1001/jamasurg.2024.0111. PMID 38446466
- [Background] El-Boghdadly K, Dhesi J, Fabb P, Levy N, Lobo DN, McKechnie A, Mustafa O, Newland-Jones P, Patel A, Pournaras DJ, Clare K, Dhatariya K. Elective peri-operative management of adults taking glucagon-like peptide-1 receptor agonists, glucose-dependent insulinotropic peptide agonists and sodium-glucose cotransporter-2 inhibitors: a multidisciplinary consensus statement: A consensus statement from the Association of Anaesthetists, Association of British Clinical Diabetologists, British Obesity and Metabolic Surgery Society, Centre for Perioperative Care, Joint British Diabetes Societies for Inpatient Care, Royal College of Anaesthetists, Society for Obesity and Bariatric Anaesthesia and UK Clinical Pharmacy Association. Anaesthesia. 2025 Apr;80(4):412-424. doi: 10.1111/anae.16541. Epub 2025 Jan 9. PMID 39781571
- [Background] Lin H, He JJ, Cai ZS, Lu ZW, Lin ZJ, Lin XZ, Huang QW. Ultrasonic evaluation of metoclopramide's effect on gastric motility in emergency trauma patients. Front Physiol. 2023 May 10;14:999736. doi: 10.3389/fphys.2023.999736. eCollection 2023. PMID 37234409
- [Background] Shakhatreh M, Jehangir A, Malik Z, Parkman HP. Metoclopramide for the treatment of diabetic gastroparesis. Expert Rev Gastroenterol Hepatol. 2019 Aug;13(8):711-721. doi: 10.1080/17474124.2019.1645594. Epub 2019 Jul 30. PMID 31314613
- [Background] Ushakumari DS, Sladen RN. ASA Consensus-based Guidance on Preoperative Management of Patients on Glucagon-like Peptide-1 Receptor Agonists. Anesthesiology. 2024 Feb 1;140(2):346-348. doi: 10.1097/ALN.0000000000004776. No abstract available. PMID 37982170
- [Background] Joshi GP. Anesthetic Considerations in Adult Patients on Glucagon-Like Peptide-1 Receptor Agonists: Gastrointestinal Focus. Anesth Analg. 2024 Jan 1;138(1):216-220. doi: 10.1213/ANE.0000000000006810. Epub 2023 Dec 15. No abstract available. PMID 37874648
- [Background] Gariani K, Putzu A. Glucagon-like peptide-1 receptor agonists in the perioperative period: Implications for the anaesthesiologist. Eur J Anaesthesiol. 2024 Mar 1;41(3):245-246. doi: 10.1097/EJA.0000000000001914. Epub 2024 Feb 2. No abstract available. PMID 38298102
- [Background] Yao H, Zhang A, Li D, Wu Y, Wang CZ, Wan JY, Yuan CS. Comparative effectiveness of GLP-1 receptor agonists on glycaemic control, body weight, and lipid profile for type 2 diabetes: systematic review and network meta-analysis. BMJ. 2024 Jan 29;384:e076410. doi: 10.1136/bmj-2023-076410. PMID 38286487
- [Background] Asai T. Editorial II: Who is at increased risk of pulmonary aspiration? Br J Anaesth. 2004 Oct;93(4):497-500. doi: 10.1093/bja/aeh234. No abstract available. PMID 15361474
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489